CLINICAL TRIAL: NCT05570552
Title: Long Term Effects of Household Air Pollution (HAP) Reduction on Cardio-pulmonary and Immune Function Outcomes - a Household Level Randomized mHealth Intervention Trial
Brief Title: 1/2- Bangladesh Center for Global Environmental and Occupational Health- Bangladesh
Acronym: GEOHealth-II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Chicago (Other); Mailman School of Public Health (Unknown); Marquette University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-22057 (2U01TW010120-06)
Record Dates: First submitted 2022-08-29; First posted 2022-10-06 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Air Pollution; mHealth Intervention; Cardiopulmonary Function; Immune Function
Keywords: Mobile based Behavioral Change Communication intervention; Household air pollution reduction; Cardiopulmonary function; Immune function; Clean fuel LPG

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth arm (Experimental): mHealth arm will receive mobile phone based behavior change communication intervention to exclusively use clean fuel LPG for domestic cooking.
  Interventions: Behavioral: mHealth based behavioral change communication intervention
- Control arm (No Intervention): Control arm will receive no mHealth based intervention.

INTERVENTIONS:
Behavioral: mHealth based behavioral change communication intervention — We will implement a mHealth based communication system. The number of text messages and push notifications that a participant receives, will be variable and will occur at least weekly (based upon their responses) or the participant opts out of receiving messages. Participant change of behavior and use of improved stoves will be monitored by tracking clicks/views of educational materials and video vignettes.
  Other Names: value sensitive design (VSD), Fogg Behavior Model (FBM), System Usability Scale (SUS)
  Arms: mHealth arm

SUMMARY:
Almost 3 billion people worldwide, including 89% people in Bangladesh, are exposed to harmful household air pollutants (HAP) emitted from combustion of biomass (wood, agricultural residue, cow dung, etc.) fuel use for cooking. While health risks associated with air-pollution have been reasonably well-studied in developed countries, there is little evidence on health benefits achievable by HAP reduction through clean fuel use, especially in low- and middle-income countries (LMICs). Earlier the investigators showed that Liquid Petroleum Gas (LPG) for 24 months, reduced personal PM2.5 exposure by 58.17 percent which induced novel changes in immune and inflammatory responses in the participants; however cardiopulmonary markers remained relatively stable in post-intervention assessment.

In this study, the investigators aim to evaluate the effects of mobile phone based (mHealth) Behavioural Change Communication (BCC) intervention on adoption and exclusive use of LPG. The investigators also aimed to observe whether long-term effects of HAP reduction can impact the subclinical measures of cardio-vascular and pulmonary dysfunction and regulate innate and inflammatory immune function among women and children in semi-rural settings in Bangladesh. The investigators will also investigate the influence of exposure to HAP on antibody response to vaccines (adaptive immunity). The BCC intervention will be provided by conducting a large household level randomized controlled trial by educational intervention using mHealth based technology. In addition, the investigators will continue following the cohort and will conduct rigorous and repeated personalized (24 hours) and area (over 5 days) assessments of PM2.5 and black carbon (BC) exposure to examine the long-term effects of HAP reduction on subclinical measures of cardio-pulmonary and immune dysfunction including effect of HAP exposure on antibody response to vaccine.

DETAILED DESCRIPTION:
Background:

Almost 3 billion people worldwide, including 89% people in Bangladesh, are exposed to harmful household air pollutants (HAP) emitted from combustion of biomass fuel (wood, agricultural residue, cow dung, etc.) used for cooking. While health risks associated with air-pollution have been reasonably well-studied in developed countries, there is little evidence on health benefits achievable by HAP reduction through clean fuel use such as Liquid Petroleum Gas, especially in low- and middle-income countries (LMICs).

Rationale: In the earlier GEOHealth (Round-I) study, the investigators have shown that LPG for 24 months, reduced personal PM2.5 exposure by 58.2 percent which induced novel changes in innate immune and inflammatory responses in women but the changes in chronic cardio-pulmonary markers were not prominent, most likely due to short duration of follow up and probably impact of ambient pollution. Moreover, sustained use of LPG could be challenging as earlier GEOHealth (Round-I) study provided the cook stove and supply of LPG free of cost. A post-completion screening showed >70% households continued using LPG albeit not exclusively. It is plausible that an intervention using mobile phone-based application can improve the exclusive use of LPG in the communities.

Hypothesis:

1. The mobile phone based (mHealth) Behavioural Change Communication (BCC) intervention can be easily incorporated in Government policy that can promote adoption, and increase exclusive use of LPG in the communities.

   The long-term effect of HAP reduction can be associated with-
2. subclinical measures of cardio-vascular and pulmonary dysfunction.
3. balanced changes in innate/ inflammatory and adaptive immune function (vaccine response).

Objectives: To evaluate

1. The effects of a scalable educational intervention (using mHealth application) on adoption and exclusive use of LPG.
2. The long-term effects of HAP reduction on subclinical measures of cardio-vascular and pulmonary dysfunction.
3. The long-term effects of HAP reduction on innate/ inflammatory immune function among women and children and to investigate the influence of HAP exposure on antibody response to vaccines (adaptive immunity).

Methods: The investigators will conduct a large household level randomized controlled trial by educational intervention using mobile phone (mHealth) based technology. In addition, the investigators will continue following the cohort and will conduct rigorous and repeated personalized (24 hours) and area-wise (over 5 days) assessments of PM2.5 and black carbon (BC) exposure to examine the long-term effects of HAP reduction on subclinical measures of cardio-pulmonary and immune dysfunction including effect of HAP exposure on antibody response to vaccine.

Outcome measures/variables: Personal and surrounding area PM2.5 and BC level will be measured at pre- and post-intervention. Lung function and lung pathology will be assessed through spirometry, Chest X-ray, and High-resolution Computed tomography of the chest (HRCT). Preclinical makers of cardiovascular diseases (CVD) will include blood pressure and EKG. Markers of metabolic dysfunction will be assesses by measuring HbA1c and fasting lipid profile. Immune function will be assessed by phenotyping of Immune cells, functional cytotoxic killer cells, oxidative stress of lymphocytes.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the previous GEOHEALTH round-I study
* Aged between 25 and 70 years
* Live in biomass-using home with traditional stoves
* Non-smoker and live with non-smokers
* Exposed to <10 µg/L of water arsenic

Exclusion Criteria:

* Known to have immune related illness or taking any prescription medication (particularly those that suppress or enhance immune function)
* Known to have any clinical events of CVD or lung disease, including stroke or coronary heart disease.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-06-20 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Personal air pollution | Pre-intervention
  Measurement of personal air pollution (PM2.5 and BC level) by personal air pollution monitoring device
Personal air pollution | Two-year post intervention
  Measurement of personal air pollution (PM2.5 and BC level) by personal air pollution monitoring device
Ambient air pollution | Pre-intervention
  Measurement of ambient air pollution (PM2.5) by ambient air monitoring device
Ambient air pollution | Two-year post intervention
  Measurement of ambient air pollution (PM2.5) by ambient air monitoring device
Lung function assessment by spirometry | Pre-intervention
  Lung function assessment by spirometry
Lung function assessment by spirometry | Two-year post intervention
  Lung function assessment by spirometry
Assessment lung pathology by chest X-ray and High-resolution Computed tomography | Pre-intervention
  Lung pathology will be assessed by chest X-ray for all participants and high-resolution Computed tomography of the chest (HRCT) will be performed in selected participants.
Assessment lung pathology by chest X-ray and High-resolution Computed tomography | Two-year post intervention
  Lung pathology will be assessed by chest X-ray for all participants and high-resolution Computed tomography of the chest (HRCT) will be performed in selected participants.
Measurement of cardiovascular disease (CVD) markers by measuring blood pressure | Pre-intervention
  Preclinical markers of CVD assessment by blood pressure
Measurement of cardiovascular disease (CVD) markers by measuring blood pressure | Two-year post intervention
  Preclinical markers of CVD assessment by blood pressure
Measurement of cardiovascular disease (CVD) markers by performing EKG | Pre-intervention
  Preclinical markers of CVD assessment by EKG
Measurement of cardiovascular disease (CVD) markers by performing EKG | Two-year post intervention
  Preclinical markers of CVD assessment by EKG
Evaluation of metabolic markers (diabetes) in blood at baseline. | Pre-intervention
  Assessment of metabolic dysfunction by measuring HbA1c
Evaluation of metabolic markers (diabetes) in blood after intervention. | Two-year post intervention
  Assessment of metabolic dysfunction by measuring HbA1c
Evaluation of metabolic markers (CVD) in blood. | Pre-intervention
  Assessment of metabolic dysfunction by measuring fasting lipid profile.
Evaluation of metabolic markers (CVD) in blood. | Two-year post intervention
  Assessment of metabolic dysfunction by measuring fasting lipid profile.
Assessment of immune function in blood cells | Pre-intervention
  Immune function will be assessed by phenotyping using flowcytometry
Assessment of immune function in blood cells | Two-year post intervention
  Immune function will be assessed by phenotyping using flowcytometry

CONTACTS AND LOCATIONS:
Locations (1):
- International Centre for Diarrhoeal Diseases Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
All data collected of the proposed study will be made fully available to any bonafide researcher. In general, the investigators will follow the data sharing plan developed and practiced by the NIH-funded grantees. Any data request by external researchers will be reviewed by the PIs and the AOC and the requested specific data will be made available to the through a secured web-based interface developed specifically for this project. In general, data will be made available six months after the manuscript reporting results from those specific sets of data are accepted for publication and all data requests will be processed within six months from the receipt of the request in writing. Any data requests with potential conflicts will be reviewed and decided by the AOC.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 6 months after manuscripts accepted for publication